CLINICAL TRIAL: NCT01822639
Title: An Open-Label, Randomized, Single Dose, Two-Way Crossover Pilot Study to Evaluate the Relative Bioavailability of One Amlodipine 5 mg Tablet and One Enalapril Maleate 20mg Tablet to a Fixed Dose Combination Tablet Formulation of Amlodipine (5 mg) and Enalapril Maleate (20 mg), in Healthy Adult Male and Female Subjects Under Fasting Conditions
Brief Title: A Fixed Dose Combination Amlodipine + Enalapril Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116798
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Hypertension
Keywords: Hypertension; enalapril maleate; healthy volunteers; amlodipine; pharmacokinetics
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Subjects in this arm will receive Treatment A in period 1 and Treatment B in period 2. Treatment A is co-administration of 5mg amlodipine tablet and 20 mg enalapril maleate tablet. Treatment B (GSK2944404) is fixed dose combination tablet of 5 mg amlodipine and 20 mg enalapril.
  Interventions: Drug: GSK2944404 FDC; Drug: Amlodipine 5 mg; Drug: Enalapril Maleate 20 mg
- Sequence 2 (Experimental): Subjects in this arm will receive Treatment B in period 1 and Treatment A in period 2. Treatment A is co-administration of 5mg amlodipine tablet and 20 mg enalapril maleate tablet. Treatment B (GSK2944404) is fixed dose combination tablet of 5 mg amlodipine and 20 mg enalapril.
  Interventions: Drug: GSK2944404 FDC; Drug: Amlodipine 5 mg; Drug: Enalapril Maleate 20 mg

INTERVENTIONS:
Drug: GSK2944404 FDC — Uncoated, round, yellow white bilayer fixed dose combination tablet containing 5 mg amlodipine and 20 mg enalapril for single dose oral administration in each period.
Drug: Amlodipine 5 mg — Emerald-shaped white 5 mg amlodipine table for single dose oral co-administration with enalapril maleate tablet in each period.
Drug: Enalapril Maleate 20 mg — Peach triangle shaped 20 mg enalapril maleate tablet for single dose oral co-administration with amlodipine in each period.

SUMMARY:
The study is designed to estimate the bioavailability of amlodipine and enalapril maleate fixed dose combination (FDC) relative to co-administration of amlodipine and enalapril maleate tablets. The rational for this study is to provide a more convenient dosing regimen for patients. This is an open-label, randomized, single dose, two-way crossover study, in which 16 healthy adult male and female subjects will be enrolled and dosed under fasting conditions. Each subject will participate in two treatment periods of 7 days each. There will be at least 14 days of wash out period between the two dosing periods and a follow-up period of up to 21 days after treatment period 2. The total duration of study will be approximately 35 days from the start of the first treatment.

ELIGIBILITY:
Inclusion Criteria

* Male or female aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator, in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) and Body Mass Index within the range 19 to 32 kg/meter squared (m^2) (inclusive).
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone > 40 milli international unit (MlU)/ milliliter (mL) and estradiol < 40 picogram/mL (<147 picomoles/liter) is confirmatory]. OR Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin test at screening or prior to dosing. Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up contact visit. OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods This criterion must be followed from the time of the first dose of study medication until the follow-up contact visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine aminotransferase, alkaline phosphatase and bilirubin <=1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Based on single or averaged QT duration corrected for heart rate (QTc) values of triplicate electrocardiograms (ECGs)obtained over a brief recording period: QTc by Fridericia's formula <450 millisecond (msec).

Exclusion Criteria Based Upon Medical Histories

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (With the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as An average weekly intake of >21 units for males or >14 units for females. In Australia one unit (=standard drink) is equivalent to 10 grams of alcohol: 270 mL of full strength beer (4.8 percent), 375 mL of mid strength beer (3.5 percent), 470mL of light beer (2.7 percent), 250 mL pre-mix full strength spirit (5 percent), 100 mL of wine (13.5 percent) and 30 mL of spirit (40 percent).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Exclusion Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immuno virus antibody.
* Pregnant females as determined by positive serum hCG test at screening or at any other time points.
* Any subject with a systolic blood pressure <95 millimeter of mercury (mmHg) or with a recent history of postural symptoms.
* Orthostatic event at screening, defined as a symptomatic event (i.e. dizziness or any pre syncope or syncope) and a reduction in systolic blood pressure of 20mmHg or more and/or a reduction in diastolic blood pressure of 10 mmHg or more for standing versus supine measurement.

Other Exclusion Criteria

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Subject is mentally or legally incapacitated.
* Positive carbon monoxide on admission to the Unit.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice (and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices) from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04-03 (Actual); Primary Completion 2013-05-24 (Actual); Study Completion 2013-05-24 (Actual)

PRIMARY OUTCOMES:
Relative oral bioavailability of GSK2944404 FDC to amlodipine and enalapril maleate tablets co-administered as assessed by composite of pharmacokinetic (PK) parameters. | PK samples will be collected at Pre-dose, 0.25, 0.5, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 36, 48, 72, 96, 120, and 144 hours post dose at each dosing session.
  PK parameters include: maximum observed concentration (Cmax) of amlodipine and enalapril in all treatments, area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC[0-t]), and area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-infinity]. Bioavailability is defined as the amount of drug available at the site of action after administration.

SECONDARY OUTCOMES:
Composite of PK parameters for enalaprilat following administration of GSK2944404 and co-administration of amlodipine and enalapril maleate as data permit. | PK samples will be collected at Pre-dose, 0.25, 0.5, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose at each dosing session.
  PK parameters include: AUC (0-infinity), AUC (0-t), Cmax, time of occurrence of Cmax (tmax), percentage of AUC (0-infinity) obtained by extrapolation (percentage AUCex), last observed quantifiable concentration (Clast), and terminal phase half-life (t1/2).
Composite of PK parameters for amlodipine and enalapril maleate following administration of GSK2944404 and co-administration of amlodipine and enalapril maleate as data permit. | PK samples will be collected at Pre-dose, 0.25, 0.5, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 36, 48, 72, 96, 120, and 144 hours post dose at each dosing session.
  PK parameters include: tmax, Clast, percentage AUCex, and t1/2.
Number of participants with adverse events (AEs) as a measure of safety and tolerability. | Up to 35 days.
  AEs will be collected from the start of Study Treatment and until the follow-up contact visit.
Vital signs measurements to assess safety and tolerability. | Up to 35 days.
  Vital signs include blood pressure and pulse rate measurement. Orthostatic (sitting in upright position) as well as supine vitals will be measured.
Absolute values and change over time of Clinical laboratory parameters to assess safety and tolerability. | Up to 35 days.
  Clinical laboratory parameters include: hematology, clinical chemistry, urinalysis and additional parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116798 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116798?search=study&study_ids=116798#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116798 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register